CLINICAL TRIAL: NCT04563104
Title: Lung Ultrasound in Procalcitonin- Guided Antibiotic Discontinuation in Ventilator Associated Pneumonia
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mona Ammar, Assistant professor, Ain Shams University
Other Study IDs: R 49 / 2020
Record Dates: First submitted 2020-09-09; First posted 2020-09-24 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2020-09

CONDITIONS: Ventilator Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Lung Ultrasound — We will evaluate the role of lung ultrasound on the duration of antibiotics, we hypothesize that ultrasound imaging may have a role, will be correlated with, procalcitonin (PCT). The created database will help in establishing conclusion and recommendations that will help to improve the antibiotics duration and decrease the resistance.

SUMMARY:
Ventilator Associated pneumonia (VAP) is associated with longer ICU length of stay, prolonged mechanical ventilation, and increased use of antimicrobials, health-care cost and mortality . Acute respiratory infections (ARIs) comprise a large and heterogeneous group of infections, including bacterial infections, viral infections, and infections of other etiologies. Early initiation of adequate antibiotic therapy is the cornerstone in the treatment. However, overuse of antibiotics and prolonged duration of antibiotic therapy in patients with bacterial ARIs in the hospital and intensive care setting is associated with increased resistance for common bacteria, high costs, and adverse drug reactions.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or greater
* Ventilator associated pneumonia (VAP) with positive sputum culture.

Exclusion Criteria:

* pregnancy,
* use of immunosuppressive agents except for steroids,
* neutropenia (white blood cell count ≤1000/mL)
* patients whose primary diagnosis was community acquired pneumonia and other source of infection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients having ventilator associated pneumonia (VAP) with positive sputum culture. VAP was considered if the onset occurred following intubation of the trachea for 48 h and the infection was absent before starting mechanical ventilation . Diagnosis of pneumonia was based on radiographic finding of pulmonary infiltrate; findings should be new and progressive and at least should satisfy two clinical criteria of the following: body temperature >38°C or <35.5°C; leukocyte count > 12,000 cells/mm3 or <4000 cells/mm3; and clinical evidence of pneumonia, such as purulent secretions and a decrease in oxygenation.
  Diagnosis of VAP was confirmed microbiologically by positive bronchial secretion cultures
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
correlation between lung ultrasound and procalcitonin. | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No